CLINICAL TRIAL: NCT00003851
Title: Evaluation of Intensive Pancreatic Proteolytic Enzyme Therapy With Ancillary Nutritional Support Versus Gemcitabine Chemotherapy in the Treatment of Inoperable Pancreatic Adenocarcinoma
Brief Title: Gemcitabine Compared With Pancreatic Enzyme Therapy Plus Specialized Diet (Gonzalez Regimen) in Treating Patients Who Have Stage II, Stage III, or Stage IV Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Approval lapse
Sponsor: Columbia University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAA8471; CPMC-IRB-8544; NCCAM; NCI-V99-1538
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Malnutrition; Pancreatic Cancer
Keywords: malnutrition; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Malnutrition; Pancreatic Neoplasms | interventions — Peptide Hydrolases; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional Arm (Active Comparator): Arm I (Nutritional Arm): Patients receive pancreatic enzymes orally every 4 hours and at meals daily on days 1-16, followed by 5 days of rest. Patients receive magnesium citrate and Papaya Plus with the pancreatic enzymes. Additionally, patients receive nutritional supplementation with vitamins, minerals, trace elements, and animal glandular products 4 times per day on days 1-16, followed by 5 days of rest. Courses repeat every 21 days until death despite relapse. Patients consume a moderate vegetarian metabolizer diet during the course of therapy, which excludes red meat, poultry, and white sugar. Coffee enemas are performed twice a day, along with skin brushing daily, skin cleansing once a week with castor oil during the first 6 months of therapy, and a salt and soda bath each week. Patients also undergo a complete liver flush and a clean sweep and purge on a rotating basis each month during the 5 days of rest.
  Interventions: Biological: proteolytic enzymes; Procedure: Gonzalez regimen
- Chemotherapy Arm (Active Comparator): Arm II (Chemotherapy Arm): Patients receive gemcitabine-based chemotherapy. Quality of life is assessed at 0, 2, 6, and 12 months and then yearly thereafter.
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: proteolytic enzymes
  Arms: Nutritional Arm
Drug: gemcitabine hydrochloride
  Arms: Chemotherapy Arm
Procedure: Gonzalez regimen
  Arms: Nutritional Arm

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Pancreatic enzymes may help kill cancer cells. It is not yet known if gemcitabine is more effective than pancreatic enzyme therapy plus specialized diet for pancreatic cancer.

PURPOSE: This clinical trial is comparing the effectiveness of gemcitabine with that of pancreatic enzyme therapy plus specialized diet (Gonzalez regimen) in treating patients who have stage II, stage III, or stage IV pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with stage II, III, or IV adenocarcinoma of the pancreas treated with gemcitabine versus intensive proteolytic enzyme therapy and adjunctive dietary and nutritional support.
* Compare the quality of life in patients treated with these regimens.

OUTLINE: This is an open-label study. Patients are stratified according to stage (II or III vs IV), performance status (0-1 vs 2) and nutritional status (well nourished or moderately malnourished vs severely malnourished). Patients are entered into 1 of 2 treatment arms at their choice:

* Arm I (Nutritional Arm): Patients receive pancreatic enzymes orally every 4 hours and at meals daily on days 1-16, followed by 5 days of rest. Patients receive magnesium citrate and Papaya Plus with the pancreatic enzymes. Additionally, patients receive nutritional supplementation with vitamins, minerals, trace elements, and animal glandular products 4 times per day on days 1-16, followed by 5 days of rest. Courses repeat every 21 days until death despite relapse. Patients consume a moderate vegetarian metabolizer diet during the course of therapy, which excludes red meat, poultry, and white sugar. Coffee enemas are performed twice a day, along with skin brushing daily, skin cleansing once a week with castor oil during the first 6 months of therapy, and a salt and soda bath each week. Patients also undergo a complete liver flush and a clean sweep and purge on a rotating basis each month during the 5 days of rest.
* Arm II (Chemotherapy Arm): Patients receive gemcitabine-based chemotherapy. Quality of life is assessed at 0, 2, 6, and 12 months and then yearly thereafter.

Patients are followed at 1, 3, 7, and 12 months and then yearly thereafter.

PROJECTED ACCRUAL: Approximately 72-90 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable primary or metastatic adenocarcinoma of the pancreas diagnosed within the past 8 weeks

  * Stage II-IV

PATIENT CHARACTERISTICS:

Age:

* 18 to physiologic 65

Performance status:

* ECOG 0-2

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.5 times normal
* SGOT or SGPT less than 1.5 times normal
* Albumin greater than 3.2 g/dL

Renal:

* Creatinine less than 1.5 times normal
* BUN less than 1.5 times normal

Other:

* Not pregnant or nursing
* HIV negative
* No other serious medical or psychiatric illness that would preclude study participation
* No serious infection
* Ability to eat solid food three meals per day
* No allergy or intolerance to pork
* No prior illicit drug addiction
* At least one year since prior daily alcohol use
* At least one year since prior cigarette use
* Must have supportive live-in spouse or other family member

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except:

  * Steroids for antiemesis, documented CNS metastases, adrenal failure, or septic shock
  * Hormonal therapy for nondisease related conditions (e.g., thyroid replacement therapy)

Radiotherapy:

* No prior radiotherapy
* Concurrent palliative radiotherapy allowed, including to a symptomatic lesion or one which may produce disability (e.g., unstable femur or CNS lesion)

Surgery:

* Greater than 1 week since prior exploratory or palliative bypass surgery
* No prior Whipple procedure or surgical procedure for curative intent

Other:

* No oral hypoglycemic agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 1999-03; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Chabot, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States

REFERENCES:
- [Result] Chabot JA, Tsai WY, Fine RL, Chen C, Kumah CK, Antman KA, Grann VR. Pancreatic proteolytic enzyme therapy compared with gemcitabine-based chemotherapy for the treatment of pancreatic cancer. J Clin Oncol. 2010 Apr 20;28(12):2058-63. doi: 10.1200/JCO.2009.22.8429. Epub 2009 Aug 17. PMID 19687327